CLINICAL TRIAL: NCT05150847
Title: The Effect of Prone Positioning on Oxygenation and Respiratory Mechanics in Patients With COVID-19 Pneumonia
Brief Title: Prone Positioning in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kazim Rollas, Intensive Care Specialist, Principal Investigator, Tepecik Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021/11-02
Record Dates: First submitted 2021-12-07; First posted 2021-12-09 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Disease 2019; ARDS; Mechanical Ventilation Pressure High
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone Positioning (Other): Patients will be ventilated in volume-controlled mode with Vt at 6 ml/kg of predicted body weight. Prone positioning will be performed over periods of 16 hours when PaO2/FiO2 was persistently lower than 150 mm Hg. Flow, volume, and airway pressure will bw measured by ventilators. Measurements of oxygenation and respiratory mechanics were performed at 5 and 15 cmH20 PEEP levels and will be repeated every season as before first period of prone positioning, before supine positioning, and again before second period of prone positioning. Total PEEP and plateau pressure will be measured by a short end-expiratory and an end-inspiratory occlusion respectively. Complete airway closure will be assessed by performing a low-flow (4 L/min) inflation( PV tool) (9). The potential for lung recruitment will be assessed by means of the R/I ratio (10).
  Interventions: Other: Oxygenation

INTERVENTIONS:
Other: Oxygenation — Oxygenation will be calculated as PaO2/ FiO2 ratio.Static compliance will be calculated as tidal volume divided driving pressure.The potential for lung recruitment will be assessed by means of the R/I ratio (10).
  Other Names: static compliance, Recruitability

SUMMARY:
Prone positioning improves oxygenation in patients with ARDS (1-3). Patients with severe ARDS due to COVID-19 are candidates for prone position. It should be started within 36-48 h and maintained 1, 3). Prone ventilationARDS based on a randomized trial that showed a mortality benefit (PROSEVA) (3).

The improvement of oxygenation occurs by making ventilation more homogeneous, limiting ventilator-associated lung injury (4-6).

Prone positioning was as effective in improving oxygenation, static respiratory system compliance (Crs) (7).

Higher PEEP should be applied when there is a high recruitability potential of the lung. This study aimed to investigate whether prone positioning changes the recruitability position of the lung.in COVID-ARDS.

DETAILED DESCRIPTION:
Prone positioning improves oxygenation in patients with ARDS (1-3). Patients with severe ARDS due to COVID-19 are candidates for prone position. It should be started within 36-48 h and maintained 1, 3). Prone ventilationARDS based on a randomized trial that showed a mortality benefit (PROSEVA) (3).

The improvement of oxygenation occurs by making ventilation more homogeneous, limiting ventilator-associated lung injury (4-6).

Prone positioning was as effective in improving oxygenation, static respiratory system compliance (Crs) (7).Higher PEEP should be applied when there is a high recruitability potential of the lung. This study aimed to investigate whether prone positioning changes the oxygenation, respiratory mechanics and recruitability position of the lung in COVID-ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with laboratory-confirmed COVID-19 admitted to the ICU
* The patients receive invasive mechanical ventilation and meet the criteria for ARDS (Berlin definition) (8), with under continuous infusion of sedatives,

Exclusion Criteria:

* Pregnancy
* Pneumothorax and or chest tube
* Chronic obstructive lung disease
* interstitial lung disease
* intraabdominal hypertension
* increase in intracranial blood pressure
* Haemodynamic unstability requiring vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-13 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | intubation + 48 hours
  PaO2/FiO2

SECONDARY OUTCOMES:
Static compliance | intubation + 48 hours
  Tidal volume divided driving pressure
Recruitability | intubation + 48 hours
  recruitment to inflation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Işıl Köse Güldoğan, Study Chair — İzmi̇r Tepeci̇k Eği̇ti̇m Ve Arştırma Hastanesi̇
Locations (1):
- Kazim Rollas, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Will be shared as the first patient included in the study
Supporting Information: Study Protocol
Time Frame: From 25 december - 3 months

REFERENCES:
- [Background] Mancebo J, Fernandez R, Blanch L, Rialp G, Gordo F, Ferrer M, Rodriguez F, Garro P, Ricart P, Vallverdu I, Gich I, Castano J, Saura P, Dominguez G, Bonet A, Albert RK. A multicenter trial of prolonged prone ventilation in severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1233-9. doi: 10.1164/rccm.200503-353OC. Epub 2006 Mar 23. PMID 16556697
- [Background] Guerin C, Gaillard S, Lemasson S, Ayzac L, Girard R, Beuret P, Palmier B, Le QV, Sirodot M, Rosselli S, Cadiergue V, Sainty JM, Barbe P, Combourieu E, Debatty D, Rouffineau J, Ezingeard E, Millet O, Guelon D, Rodriguez L, Martin O, Renault A, Sibille JP, Kaidomar M. Effects of systematic prone positioning in hypoxemic acute respiratory failure: a randomized controlled trial. JAMA. 2004 Nov 17;292(19):2379-87. doi: 10.1001/jama.292.19.2379. PMID 15547166
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Lai-Fook SJ, Rodarte JR. Pleural pressure distribution and its relationship to lung volume and interstitial pressure. J Appl Physiol (1985). 1991 Mar;70(3):967-78. doi: 10.1152/jappl.1991.70.3.967. PMID 2033012
- [Background] Cornejo RA, Diaz JC, Tobar EA, Bruhn AR, Ramos CA, Gonzalez RA, Repetto CA, Romero CM, Galvez LR, Llanos O, Arellano DH, Neira WR, Diaz GA, Zamorano AJ, Pereira GL. Effects of prone positioning on lung protection in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2013 Aug 15;188(4):440-8. doi: 10.1164/rccm.201207-1279OC. PMID 23348974
- [Background] Douglas WW, Rehder K, Beynen FM, Sessler AD, Marsh HM. Improved oxygenation in patients with acute respiratory failure: the prone position. Am Rev Respir Dis. 1977 Apr;115(4):559-66. doi: 10.1164/arrd.1977.115.4.559. PMID 322557
- [Background] Park J, Lee HY, Lee J, Lee SM. Effect of prone positioning on oxygenation and static respiratory system compliance in COVID-19 ARDS vs. non-COVID ARDS. Respir Res. 2021 Aug 6;22(1):220. doi: 10.1186/s12931-021-01819-4. PMID 34362368
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Chen L, Del Sorbo L, Grieco DL, Shklar O, Junhasavasdikul D, Telias I, Fan E, Brochard L. Airway Closure in Acute Respiratory Distress Syndrome: An Underestimated and Misinterpreted Phenomenon. Am J Respir Crit Care Med. 2018 Jan 1;197(1):132-136. doi: 10.1164/rccm.201702-0388LE. No abstract available. PMID 28557528
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Derived] Emgin O, Rollas K, Yeniay H, Elve R, Guldogan IK. Effect of the prone position on recruitability in acute respiratory distress syndrome due to COVID-19 pneumonia. Rev Assoc Med Bras (1992). 2023 May 19;69(5):e20221120. doi: 10.1590/1806-9282.20221120. eCollection 2023. PMID 37222316